CLINICAL TRIAL: NCT02263105
Title: Efficacy and Tolerability of Cisplatin Plus Alternating Weekly Temozolomide in Recurrent High-grade Gliomas: A Single-arm Prospective Phase II Clinical Study
Brief Title: Efficacy and Tolerability of Cisplatin Plus Alternating Weekly Temozolomide in Recurrent High-grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhang Zhenyu, M.D., Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT001; Huashan H (Other: Huashan H)
Record Dates: First submitted 2014-09-28; First posted 2014-10-13 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: High-grade Gliomas
Keywords: recurrent high-grade gliomas; cisplatin (CDDP); temozolomide (TMZ)
MeSH Terms: interventions — Temozolomide

ARMS (1):
- CDDP plus Temozolomide (Experimental): Patients were treated with CDDP and TMZ. CDDP was administered iv from Day 1 to 3 with everyday dose of 30mg. TMZ was orally administered from Day 1 to 7 and Day 15 to 21, with everyday dose of 125mg/m2 (Level 2). The period of one chemotherapy cycle is 28 days. TMZ dose levels were listed in Table 1.
  Table 1 TMZ dose levels Dose levels Daily TMZ dose( mg/m2/d ) TMZ dose per cycle(mg/m2)
  1. 150 2100
  2. 125 1750
  3. 100 1400
  4. 75 1050
  Interventions: Drug: CDDP; Drug: Temozolomide

INTERVENTIONS:
Drug: CDDP
Drug: Temozolomide — If hematologic and nonhematologic toxicity assessed according to the Common Terminology Criteria for Adverse Events (CTCAE; version 4.0) from the previous cycle had been grade 0 or 1, then TMZ dose escalation to was allowed to the maximum of 150 mg/m2. If grade 4 hematologic toxicity or grade 3 nonhematologic toxicity had occurred, then TMZ dose was reduced in 25 mg/m2 steps. If grade 4 nonhematologic toxicity occurred, patient treatment was halted. If grade 4 hematologic toxicity or grade 3 nonhematologic toxicity continued when TMZ dose was in the minimum of 75 mg/m2, patient treatment was halted.

SUMMARY:
Currently, the prognosis of recurrent high-grade gliomas is still dismal with no standard treatment protocol established. Cisplatin (CDDP), recommended by National Comprehensive Cancer Network (NCCN) as a chemotherapeutic agent in salvage treatment for recurrent high-grade gliomas, was shown to reduce O6-alkylguanine DNA-alkyl transferase (AGAT) activity and potentially capable of enhancing the antitumor effects of temozolomide (TMZ). Compared to the standard 5-day TMZ regimen, alternating weekly regimen that deliver more prolonged exposure of TMZ may lead to higher cumulative doses, and may deplete more O6-methylguanine DNA methyltransferase (MGMT), thus reducing the resistance of tumor cells to TMZ.

The investigators therefore initiate a single-arm Phase II study to evaluate the efficacy and tolerability of CDDP plus alternating weekly TMZ regimen in patients with recurrent high-grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary tumor as high-grade gliomas (WHO III or IV)
* All patients should complete radiation therapy for primary gliomas.
* MRI showed unequivocal evidence of tumor recurrence or progression.
* The time to be enrolled should be more than 90 days after the radiation therapy.
* Written informed consent
* Eastern Cooperative Oncology Group(ECOG) score: 0-2
* The patients with recurrent gliomas were treated without dose-dense TMZ therapy before enrollment.
* Surgical interventions for recurrent gliomas are permitted and patients with no residual tumor are permitted

Exclusion Criteria:

* Abnormal function of liver or renal (value more than 1.5 fold normal upper limit)
* Blood routing: Hb < 90g/L, absolute neutrophil count≤1.5*10^9/L, platelet < 100*10^9/L
* Pregnant or lactating women
* Allergic to administered drugs
* Radiation therapy in the previous 90 days before enrollment
* The patients with recurrent gliomas were treated with dose-dense TMZ therapy before enrollment.
* Acute infection in need of antibiotics intravenously
* Participation in other clinical trials in the 90 days before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | at 6 months

SECONDARY OUTCOMES:
overall survival(OS) | at 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Qin, MD, Study Chair — Huashan Hospital; Ying Mao, MD, Principal Investigator — Huashan Hospital; Yu Yao, MD, Principal Investigator — Huashan Hospital; ZhenYu Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China